CLINICAL TRIAL: NCT05903586
Title: Vascular Changes in Patients With Aotic Isthmus Stenosis After Interventional Therapy Using Ballon Angioplasty or Stent Implantation
Brief Title: Vascular Changes in Patients With Aotic Isthmus Stenosis After Interventional Therapy
Acronym: ISTHA
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Agnes Bosch, Dr. med. Agnes Bosch, Principal Investigator, University of Erlangen-Nürnberg Medical School
Other Study IDs: ISTHA
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Aortic Isthmus Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This controlled clinical study investigates arterial blood pressure and vascular remodling before and 4 weeks after catheter interventional treatment of re-stenosis of the aortic isthmus (Recoarctatio Aortae).

DETAILED DESCRIPTION:
Patients with treated aortic isthmus stenosis during their first year of life often develop a Recoarctatio Aortae (re-stenosis of the aortic isthmus) in the long term followed by arterial hypertension. The Recoarctatio Aortae can be treated during a cather intervention by balloon dilatation or stent implantation. Patients with arterial hypertension often develop vascular remodeling with increased central systolic blood pressure and increased pulse pressure. Vascular remodling predics cardiovascular events and increases mortality. Vascular remodeling can be assessed non-invasively by using scanning laser doppler flowmetry (SLDF)), pulse wave analysis and measurement of flow-dependent vasodilation. In this controlled clinical study we investigate arterial blood pressure and vascular remodling before and 4 weeks after catheter interventional treatment of Recoarctatio Aortae.

ELIGIBILITY:
Inclusion Criteria:

* male and female persons with Recoarctatio Aortae and planned interventional therapy (balloon dilatation or stent implantation)
* adequate contraceptive methods in females with childbearing potential

Exclusion Criteria:

* other secondary causes for hypertension
* treatment resistent arterial hypertension or uncontrolled hypertension (office BP ≥ 180/110 mmHg)
* history of hypertensive enzephalopathy or intracerebral bleeding
* diabetes mellitus
* cataract
* known renal, respiratory, hepatic, gastrointestinal, endocrine, metabolic, immunolic, hematologic, oncologic, neurologic or psychiatric diseases besides the diagnosis of artoic isthmus stenosis
* one of the following diseases or conditions during the last 6 months: myocardial infaction, instable angina pectoris, cardiac insufficiency
* pregnant or lactating woman or inadequate contraception (pearl-index ≥ 1%)
* participation in another clinical study
* drug or medication abuse
* inadequate adherence or other condition preventing the patient from study participation (in the eyes of the treating physician)

Ages: 12 Years to 99 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Recoarctatio Aortae and planned interventional therapy (balloon dilatation or stent implantation)
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
change in central systolic blood pressure (BP) (mmHg) measured using pulse wave analysis | 4 weeks
  change in central systolic blood pressure (BP) (mmHg) between baseline and 4 weeks post intervention

SECONDARY OUTCOMES:
change in central diastolic blood pressure (BP) (mmHg) measured using pulse wave analysis | 4 weeks
  change in central diastolic blood pressure (BP) (mmHg) between baseline and 4 weeks post intervention
change in central pulse pressure measured (mmHg) using pulse wave analysis | 4 weeks
  change in central pulse pressure (mmHg) between baseline and 4 weeks post intervention
change in augmentation index (-) measured using pulse wave analysis | 4 weeks
  change in augmentation index (-) between baseline and 4 weeks post intervention
change in pulse wave velocity (m/s) | 4 weeks
  change in pulse wave velocity (m/s) between baseline and 4 weeks post intervention
change in systolic and diastolic office BP (mmHg) | 4 weeks
  change in systolic and diastolic office BP (mmHg) between baseline and 4 weeks post intervention
change in systolic and diastolic 24 hour ambulatory BP (mmHg) | 4 weeks
  change in systolic and diastolic 24 hour ambulatory BP (mmHg) between baseline and 4 weeks post intervention
change in retinal arteriolar wall to lumen ratio (-) measured using Scanning Laser Doppler Flowmetry | 4 weeks
  change in retinal arteriolar wall to lumen ratio between baseline and 4 weeks post intervention
change in retinal capillary flow (AU) measured using Scanning Laser Doppler Flowmetry | 4 weeks
  change in retinal capillary flow (AU) between baseline and 4 weeks post intervention
change in retinal capillary density measured using Scanning Laser Doppler Flowmetry | 4 weeks
  change in retinal capillary density between baseline and 4 weeks post intervention
change in flow dependent vasodilation measured using the Unex Device | 4 weeks
  change in flow dependent vasodilation between baseline and 4 weeks post intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Center, Department of Nephrology and Hypertension, University Hospital Erlangen, Erlangen, Germany